CLINICAL TRIAL: NCT00580606
Title: Sublingual Immunotherapy for Peanut Allergy: A Randomized, Double-Blind, Placebo-Controlled, Phase I/II Pilot Study With a Whole Peanut Extract
Brief Title: A Randomized, Double-Blind Placebo-Controlled Peanut Sublingual Immunotherapy Trial
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Consortium of Food Allergy Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: DAIT CoFAR4
Record Dates: First submitted 2007-12-18; First posted 2007-12-25 (Estimated); Results first posted 2012-10-30 (Estimated); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Food Hypersensitivity; Hypersensitivity; Immediate Hypersensitivity; Peanut Hypersensitivity
Keywords: Food Allergy; Peanut Allergy; Sublingual Immunotherapy
MeSH Terms: conditions — Food Hypersensitivity; Hypersensitivity; Hypersensitivity, Immediate; Peanut Hypersensitivity | interventions — Glycerol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Low Dose Peanut SLIT (Double Blind to Open Label) (Experimental): Subjects ingest peanut protein (glycerinated peanut allergenic extract) daily starting with 0.000165 mcg, followed by a build-up phase (escalating peanut doses every 2 weeks, achieving maintenance dose by 36 weeks). Thereafter, subjects are on a maximally tolerated maintenance dose (165 mcg to 1,386 mcg) for >= 8 weeks. After Week 44, subjects are given a 5,000 mg Oral Food Challenge (OFC) using peanut powder. Subjects/study staff are unblinded following this OFC and continue on an open label peanut protein maintenance dose of 1,386 mcg/day or may attempt escalation up to this dose. Subjects who at the Week 116 OFC are unable to consume >= 5,000 mg peanut powder or 10-fold the amount of peanut powder compared to the baseline OFC will discontinue study therapy. SLIT=Sublingual Immunotherapy.
  Interventions: Drug: Glycerinated peanut allergenic extract
- Placebo (DB) Crossed Over to High Dose Peanut SLIT (OL) (Placebo Comparator): Subjects ingest placebo (glycerin) daily beginning with a dose of 0.000165 mcg, followed by a build-up phase (escalating placebo doses every 2 weeks, achieving a maintenance dose by 36 weeks). Thereafter, subjects are on a maximally tolerated maintenance dose (165 mcg to 1,386 mcg) for >= 8 weeks. After Week 44, subjects are given a 5,000 mg Oral Food Challenge (OFC) using peanut powder. Subjects/study staff are unblinded following this OFC and subjects no longer receive placebo dosing but are crossed over and receive open label high dose peanut SLIT; the study procedures and schedule are the same as for the Low Dose Peanut SLIT group, the only difference is the maximum maintenance dose is almost 3-fold higher at 3,696 mcg/day. DB=Double Blind, SLIT=Sublingual Immunotherapy, OL=Open Label.
  Interventions: Drug: Placebo for peanut extract (glycerin)

INTERVENTIONS:
Drug: Glycerinated peanut allergenic extract — Glycerinated peanut extract delivered sublingually.
  Other Names: Peanut SLIT
  Arms: Low Dose Peanut SLIT (Double Blind to Open Label)
Drug: Placebo for peanut extract (glycerin) — Placebo (glycerin) delivered sublingually.
  Other Names: Placebo
  Arms: Placebo (DB) Crossed Over to High Dose Peanut SLIT (OL)

SUMMARY:
The purpose of this study is to evaluate the safety and immune response to daily sublingual (under the tongue) immunotherapy (SLIT) with peanut extract in adults and children with peanut allergies.

DETAILED DESCRIPTION:
Peanut allergy is a common ailment in the United States. Research suggests that the prevalence of peanut allergy in the United States has doubled over the last 5 years. Currently, the only effective treatment for peanut allergy is a peanut-free diet and quick access to self-injectable epinephrine in the event of peanut exposure. The sublingual route is a potential method to administer immunotherapy for the treatment of food allergies. The intent of this study is to induce desensitization and eventually tolerance to peanut protein and evaluate the safety and immunologic effects of daily sublingual immunotherapy (SLIT) for individuals with peanut allergy. The trial will enroll 40 participants. After the first 10 participants between the ages of 18 and 40 are enrolled, safety information will be reviewed. If there are no safety concerns, the study will continue to enroll the remaining participants between the ages of 12 and 40.

This clinical trial will last 172 to 216 weeks. Participants will be randomly assigned to receive peanut SLIT or placebo SLIT. All participants will have an entry oral food challenge (OFC). The treatment group will receive gradual dosing escalations of peanut SLIT and maintenance therapy over a 44-week period, followed by another OFC. Following the OFC, participants will be unblinded, and the placebo group will receive peanut SLIT escalated to a higher maximum dose than the first treatment group. Maintenance therapy will continue for both groups for more than 2 years.

Study visits will occur every 2 weeks during dosing escalations of peanut SLIT, followed by visits gradually spacing out during maintenance to every 12 weeks. At selected visits, a physical examination, skin prick tests, blood and urine collection, and atopic dermatitis and asthma evaluations will occur. Approximately 6 OFCs will be administered to each participant throughout the course of the study. Additionally, 10 participants will be enrolled as control participants who will not receive any study therapy and will only have blood drawn at 3 visits throughout the course of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Physician-diagnosed peanut allergy OR convincing clinical history of peanut allergy
* Reacts to a cumulative dose of 2,000 mg or less of peanut powder
* Positive peanut allergy skin prick test OR detectable serum peanut-specific IgE level
* Willing to use an acceptable method of contraception for the duration of the study
* Ability to perform spirometry maneuver in accordance with the American Thoracic Society guidelines

Exclusion Criteria:

* History of severe anaphylaxis to peanut
* Currently participating in a study using a new investigational new drug
* Participation in any interventional study for the treatment of food allergy in the 12 months prior to study entry
* Allergic to placebo ingredients (glycerin or oat flour) OR reacts to any dose of placebo during study entry oral food challenge (OFC)
* Currently in a buildup phase of any allergy immunotherapy
* Poor control of atopic dermatitis
* Moderate or severe asthma despite therapy
* Current treatment with greater than medium daily doses of inhaled corticosteroids
* Use of steroid medications
* Use of omalizumab or other nontraditional forms of allergen immunomodulatory therapy (not including corticosteroids) or biologic therapy in the 12 months prior to study entry
* Use of beta blockers, angiotensin-converting enzyme inhibitors, angiotensin-receptor blockers, or calcium channel blockers
* Inability to discontinue antihistamines for skin testing and OFCs
* History of ischemic cardiovascular disease
* History of alcohol or drug abuse
* Other significant medical conditions that, in the opinion of the investigator, prevent participation in the study
* Previous intubation due to allergies or asthma
* Uncontrolled high blood pressure
* Pregnancy or breastfeeding

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2007-12; Primary Completion 2010-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wesley Burks, MD, Study Chair — Duke University; David Fleischer, MD, Study Chair — National Jewish Health; Hugh A. Sampson, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Stacie Jones, MD, Principal Investigator — Arkansas Children's Hospital Research Institute; Robert Wood, MD, Principal Investigator — Johns Hopkins University
Locations (5):
- United States (5):
  - University of Arkansas, Little Rock, Arkansas
  - National Jewish Medical and Research Center, Denver, Colorado
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Mount Sinai School of Medicine, New York, New York
  - University of North Carolina, Durham, North Carolina

REFERENCES:
- [Background] de Leon MP, Rolland JM, O'Hehir RE. The peanut allergy epidemic: allergen molecular characterisation and prospects for specific therapy. Expert Rev Mol Med. 2007 Jan 9;9(1):1-18. doi: 10.1017/S1462399407000208. PMID 17210088
- [Background] Enrique E, Cistero-Bahima A. Specific immunotherapy for food allergy: basic principles and clinical aspects. Curr Opin Allergy Clin Immunol. 2006 Dec;6(6):466-9. doi: 10.1097/01.all.0000246618.41871.a4. PMID 17088653
- [Background] Sicherer SH, Sampson HA. Peanut allergy: emerging concepts and approaches for an apparent epidemic. J Allergy Clin Immunol. 2007 Sep;120(3):491-503; quiz 504-5. doi: 10.1016/j.jaci.2007.07.015. Epub 2007 Aug 8. PMID 17689596
- [Result] Fleischer DM, Burks AW, Vickery BP, Scurlock AM, Wood RA, Jones SM, Sicherer SH, Liu AH, Stablein D, Henning AK, Mayer L, Lindblad R, Plaut M, Sampson HA; Consortium of Food Allergy Research (CoFAR). Sublingual immunotherapy for peanut allergy: a randomized, double-blind, placebo-controlled multicenter trial. J Allergy Clin Immunol. 2013 Jan;131(1):119-27.e1-7. doi: 10.1016/j.jaci.2012.11.011. PMID 23265698
- [Result] Burks AW, Wood RA, Jones SM, Sicherer SH, Fleischer DM, Scurlock AM, Vickery BP, Liu AH, Henning AK, Lindblad R, Dawson P, Plaut M, Sampson HA; Consortium of Food Allergy Research. Sublingual immunotherapy for peanut allergy: Long-term follow-up of a randomized multicenter trial. J Allergy Clin Immunol. 2015 May;135(5):1240-8.e1-3. doi: 10.1016/j.jaci.2014.12.1917. Epub 2015 Feb 3. PMID 25656999
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: Main Areas of Focus: Consortium of Food Allergy Research (CoFAR) — https://www.niaid.nih.gov/research/consortium-food-allergy-research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place at five university-based medical centers in the United States (Mt. Sinai School of Medicine, Johns Hopkins University, Duke University, National Jewish Medical Center, University of Arkansas Children's Hospital from April 2008 to January 2010.
Period: Double Blind (DB)
Arm/Group | Low Dose Peanut SLIT (Double Blind to Open Label) | Placebo (DB) Crossed Over to High Dose Peanut SLIT (OL)
Started | 20 | 20
Had Week 44 Oral Food Challenge | 18 | 19
Completed | 20 (Completed: Participants who were assessed for the primary outcome measure.) | 20 (Completed: Participants who were assessed for the primary outcome measure.)
Not Completed | 0 | 0
Period: Open Label (OL)
Arm/Group | Low Dose Peanut SLIT (Double Blind to Open Label) | Placebo (DB) Crossed Over to High Dose Peanut SLIT (OL)
Started | 18 (2 participants discontinued dosing before Open Label (OL) period.) | 17 (1 participant discontinued dosing before OL period; 2 passed Week 44 OFC & ineligible to crossover.)
Had Week 44 Oral Food Challenge | 0 (The Week 44 OFC for Low Dose Peanut SLIT was done at the end of the DB Period, not the OL period.) | 12 (After 44 weeks of OL high dose SLIT; 1 additional participant declined Week 44 OFC in OL period.)
Had Week 68 Oral Food Challenge | 15 | 12
Had Week 116 Oral Food Challenge | 13 | 6
Had Week 164 Oral Food Challenge | 9 | 5
Had Week 172 Oral Food Challenge | 2 | 2
Completed | 9 (Completed dosing & final Wk 164 desensitization OFC & Wk 172 tolerance OFC (if passed Wk 164 OFC).) | 5 (Completed dosing & final Wk 164 desensitization OFC & Wk 172 tolerance OFC (if passed Wk 164 OFC).)
Not Completed | 9 | 12
Not completed — Lack of Efficacy at Week 116 OFC | 2 | 1
Not completed — Withdrawal by Subject | 4 | 6
Not completed — Dosing Symptoms | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Pregnancy | 0 | 1
Not completed — Non-compliance | 2 | 0
Not completed — Physician Decision | 1 | 1
Not completed — Needed Prohibited Medication | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Dose Peanut SLIT (Double Blind to Open Label) | Placebo (DB) Crossed Over to High Dose Peanut SLIT (OL) | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 15 | 15 | 30
  Between 18 and 65 years | 5 | 5 | 10
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 17.2 (7.6) | 16.5 (3.5) | 16.8 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 13 | 14 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 20 | 20 | 40
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 17 | 19 | 36
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40
Atopic Dermatitis Total Score [Mean (Standard Deviation); unit: Scores on a scale] — The Atopic Dermatitis Total Score is scored on a 10 point scale of 0 to 9 where a higher score indicates increasing severity of atopic dermatitis. This score is a combination of three scores that range from 0 to 3 in the following areas: body surface area score, disease course, and disease intensity.
  Scores on a scale | 1.1 (1.7) | 0.9 (1.6) | 1.0 (1.6)
Total IgE [Mean (Standard Deviation); unit: kU/L] — Total amount of serum immunoglobulin E. Individuals who are not allergic may have a total IgE as high as 304 kU/L.
  kU/L | 407.8 (254.1) | 330.5 (305.0) | 369.1 (279.9)
Peanut IgE [Mean (Standard Deviation); unit: kUA/L] — Amount of serum peanut-specific immunoglobulin E. Individuals with a peanut IgE of <0.35 kUA/L are considered not to be sensitized to peanut.
  kUA/L | 33.6 (38.1) | 47.1 (58.0) | 40.4 (48.9)
Peanut Skin Prick Test Score [Mean (Standard Deviation); unit: mm] — This score is calculated by subtracting the size of the saline wheal (in mm) from the size of the peanut wheal (in mm) observed for a skin prick test. Individuals with a peanut skin prick test score of < 3 mm are considered to have a negative result. 1 subject in the Placebo group did not have a value for this measure.
  mm | 14.0 (6.9) | 12.4 (4.6) | 13.2 (5.9)
Age at Initial Peanut Allergic Reaction [Mean (Standard Deviation); unit: years] — Two subjects in the Placebo group did not have a value for this measure.
  years | 4.6 (6.9) | 1.9 (1.5) | 3.3 (5.2)

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants Who Successfully Consumed 5,000 mg of Peanut Powder or at Least a 10-fold Increase in the Amount of Peanut Powder Compared to Their Baseline Oral Food Challenge
Description: Desensitization Assessment: Participants who successfully consumed without dose-limiting symptoms 5,000 mg of peanut powder or at least a 10-fold increase in the amount of peanut powder compared to their baseline oral food challenge during a double-blind placebo-controlled oral food challenge were counted as successes.
Time Frame: Week 44 (Double Blind Period)
Population: The intention to treat (ITT) population was used which included all subjects randomized to double-blind treatment.
Measure: Number; unit: Percentage of participants
Groups:
- Low Dose Peanut SLIT (Double Blind): Subjects ingest peanut protein (glycerinated peanut allergenic extract) daily starting with 0.000165 mcg, followed by a build-up phase (escalating peanut doses every 2 weeks, achieving maintenance dose by 36 weeks). Thereafter, subjects are on a maximally tolerated maintenance dose (165 mcg to 1,386 mcg) for >= 8 weeks. After Week 44, subjects are given a 5,000 mg Oral Food Challenge (OFC) using peanut powder. Subjects/study staff are unblinded following this OFC and continue on an open label peanut protein maintenance dose of 1,386 mcg/day or may attempt escalation up to this dose. SLIT=Sublingual Immunotherapy, mcg=microgram
- Placebo (Double Blind): Subjects ingest placebo (glycerin) daily beginning with a dose of 0.000165 mcg, followed by a build-up phase (escalating placebo doses every 2 weeks, achieving a maintenance dose by 36 weeks). Thereafter, subjects are on a maximally tolerated maintenance dose (165 mcg to 1,386 mcg) for >= 8 weeks. After Week 44, subjects are given a 5,000 mg Oral Food Challenge (OFC) using peanut powder. Subjects/study staff are unblinded following this OFC and subjects no longer receive placebo dosing but are crossed over into the High Dose Peanut SLIT Crossover (Open Label) group. SLIT=Sublingual Immunotherapy, mcg=microgram
Arm/Group | Low Dose Peanut SLIT (Double Blind) | Placebo (Double Blind)
Number analyzed (Participants) | 20 | 20
Percentage of participants | 70 | 15
Statistical Analysis 1: Comparison: Low Dose Peanut SLIT (Double Blind) vs Placebo (Double Blind); Number of participants who successfully consumed 5,000 mg of peanut powder or at least a 10-fold increase in the amount of peanut powder compared to their baseline OFC was compared using Barnard's Statistic with the null hypothesis that there was no difference between treatment groups; Test type: Superiority or Other; p < 0.001, Barnard's Statistic — No adjustments were made to the p-value; The a priori threshold for statistical significance is 0.05; Risk Difference (RD) = 55, 95% CI 2-sided [22.2 to 77.6]

2. Secondary Outcome: Percent of Participants Who Achieved a Maintenance Dose of 1,386 mcg
Description: During the build-up phase, escalation was to occur every 2 weeks until the 1,386 mcg maintenance dose was reached. The maximum time allowed for the build-up phase was 36 weeks; the dose achieved by 36 weeks was considered the maintenance dose.
Time Frame: Week 44 (Double Blind Period)
Population: The intention to treat (ITT) population was used which included all subjects randomized to double-blind treatment.
Measure: Number; unit: Percentage of participants
Groups:
- Low Dose Peanut SLIT (Double Blind): Subjects ingest peanut protein (glycerinated peanut allergenic extract) daily starting with 0.000165 mcg, followed by a build-up phase (escalating peanut doses every 2 weeks, achieving maintenance dose by 36 weeks). Thereafter, subjects are on a maximally tolerated maintenance dose (165 mcg to 1,386 mcg) for >= 8 weeks. After Week 44, subjects are given a 5,000 mg Oral Food Challenge (OFC) using peanut powder. Subjects/study staff are unblinded following this OFC and continue on an open label peanut protein maintenance dose of 1,386 mcg/day or may attempt escalation up to this dose. SLIT=Sublingual Immunotherapy
- Placebo (Double Blind): Subjects ingest placebo (glycerin) daily beginning with a dose of 0.000165 mcg, followed by a build-up phase (escalating placebo doses every 2 weeks, achieving a maintenance dose by 36 weeks). Thereafter, subjects are on a maximally tolerated maintenance dose (165 mcg to 1,386 mcg) for >= 8 weeks. After Week 44, subjects are given a 5,000 mg Oral Food Challenge (OFC) using peanut powder. Subjects/study staff are unblinded following this OFC and subjects no longer receive placebo dosing but are crossed over into the High Dose Peanut SLIT Crossover (Open Label) group. SLIT=Sublingual Immunotherapy
Arm/Group | Low Dose Peanut SLIT (Double Blind) | Placebo (Double Blind)
Number analyzed (Participants) | 20 | 20
Percentage of participants | 85.0 | 95.0

3. Secondary Outcome: Percent of Crossover Participants Who Successfully Consumed 5,000 mg of Peanut Powder or at Least a 10-fold Increase in the Amount of Peanut Powder Compared to Their Baseline Oral Food Challenge After 44 Weeks of Open Label Peanut Protein Consumption
Description: as for outcome 1
Time Frame: Week 44 after initiating crossover open label peanut protein consumption
Population: Subjects in the Placebo group during the double-blind period who crossed over to open label high dose peanut sublingual immunotherapy were included except for 1 subject who refused the crossover Week 44 OFC and could not be evaluated. 4 subjects who discontinued dosing prior to the crossover Week 44 OFC were counted as failures.
Measure: Number; unit: Percentage of participants
Groups:
- High Dose Peanut SLIT Crossover (Open Label): Subjects ingest open label peanut protein (glycerinated peanut allergenic extract) daily beginning with a dose of 0.000165 mcg, followed by a build-up phase (escalating peanut doses every 2 weeks, achieving a maintenance dose by 36 weeks). Thereafter, subjects are on a maximally tolerated maintenance dose (165 mcg to 3,696 mcg) for >= 8 weeks. After Week 44 of open label therapy, subjects either continue on their peanut protein maintenance dose of 3,696 mcg per day or are allowed to attempt escalation up to this dose. Subjects who at their Week 116 Oral Food Challenge (OFC) are not able to consume at least 5,000 mg of peanut powder or 10-fold the amount of peanut powder compared to their baseline OFC will discontinue study therapy.
Arm/Group | High Dose Peanut SLIT Crossover (Open Label)
Number analyzed (Participants) | 16
Percentage of participants | 43.8

4. Secondary Outcome: Percent of Crossover Participants Who Achieved an Open Label Peanut Protein Consumption Maintenance Dose of 3,696 mcg
Description: During the build-up phase, escalation was to occur every 2 weeks until the 3,696 mcg maintenance dose was reached. The maximum time allowed for the build-up phase was 36 weeks; the dose achieved by 36 weeks was considered the maintenance dose.
Time Frame: Week 44 after initiating crossover open label peanut protein consumption
Population: All subjects in the Placebo group during the double-blind period who crossed over to open label high dose peanut sublingual immunotherapy were included.
Measure: Number; unit: Percentage of participants
Arm/Group | High Dose Peanut SLIT Crossover (Open Label)
Number analyzed (Participants) | 17
Percentage of participants | 88.2

5. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: This study graded the severity of Adverse Events experienced by participants according to the criteria set forth in the National Cancer Institute's Common Terminology Criteria for Adverse Events Version 3.
Time Frame: Baseline through Week 44 (Double Blind Period)
Population: The intention to treat (ITT) population was used which included all subjects randomized to double-blind treatment.
Measure: Number; unit: participants
Arm/Group | Low Dose Peanut SLIT (Double Blind) | Placebo (Double Blind)
Number analyzed (Participants) | 20 | 20
participants | 1 | 0

6. Secondary Outcome: Number of Crossover Participants With Serious Adverse Events (SAEs) During 44 Weeks of Open Label Peanut Protein Consumption
Description: All subjects who were in the Placebo group during the double-blind phase of the study who initiated crossover peanut sublingual immunotherapy during the open label phase of the study will be included.
Time Frame: Initiation of open label peanut protein study therapy through Week 44 of open label peanut protein consumption
Population: All subjects who were in the Placebo group during the double-blind phase of the study who initiated crossover peanut sublingual immunotherapy during the open label phase of the study will be included.
Measure: Number; unit: participants
Arm/Group | High Dose Peanut SLIT Crossover (Open Label)
Number analyzed (Participants) | 17
participants | 0

7. Secondary Outcome: Percent of Participants Who Successfully Consumed 10,000 mg of Peanut Powder
Description: Tolerance Assessment: Participants who successfully consumed without dose-limiting symptoms 10,000 mg of peanut powder during a double-blind placebo-controlled oral food challenge were then given an open feeding of peanut butter and those who successfully consumed the open feeding were counted as successes.
Time Frame: Approximately 8 weeks after discontinuing study therapy after 3 years on maintenance study therapy
Population: All subjects randomized to the Low Dose Peanut SLIT group and all subjects randomized to the Placebo group who crossed over to open label high dose peanut sublingual immunotherapy were included.
Measure: Number; unit: percentage of participants
Arm/Group | Low Dose Peanut SLIT (Double Blind to Open Label) | Placebo (DB) Crossed Over to High Dose Peanut SLIT (OL)
Number analyzed (Participants) | 20 | 17
percentage of participants | 10.0 | 11.8

ADVERSE EVENTS:
Time Frame: Baseline through 44 weeks of study therapy
Description: This study graded the severity of Adverse Events experienced by participants according to the criteria set forth in the National Cancer Institute's Common Terminology Criteria for Adverse Events Version 3.
Groups:
- Low Dose Peanut SLIT Before Week 44 OFC (Double Blind): Subjects ingest peanut protein (glycerinated peanut allergenic extract) daily starting with 0.000165 mcg, followed by a build-up phase (escalating peanut doses every 2 weeks, achieving maintenance dose by 36 weeks). Thereafter, subjects are on a maximally tolerated maintenance dose (165 mcg to 1,386 mcg) for >= 8 weeks. After Week 44, subjects are given a 5,000 mg Oral Food Challenge (OFC) using peanut powder. Subjects/study staff are unblinded following this OFC and subjects continue on an open label peanut protein maintenance dose of 1,386 mcg/day or may attempt escalation up to this dose. SLIT=Sublingual Immunotherapy
- Placebo Before Week 44 OFC (Double Blind): Subjects ingest placebo (glycerin) daily beginning with a dose of 0.000165 mcg, followed by a build-up phase (escalating placebo doses every 2 weeks, achieving a maintenance dose by 36 weeks). Thereafter, subjects are on a maximally tolerated maintenance dose (165 mcg to 1,386 mcg) for >= 8 weeks. After Week 44, subjects are given a 5,000 mg Oral Food Challenge (OFC) using peanut powder. Subjects/study staff are unblinded following this OFC and subjects no longer receive placebo dosing but are crossed over into the High Dose Peanut SLIT Crossover (Open Label) group. SLIT=Sublingual Immunotherapy
- High Dose Peanut SLIT Crossover Before Wk44 Crossover OFC (OL): Subjects ingest open label peanut protein (glycerinated peanut allergenic extract) daily beginning with a dose of 0.000165 mcg, followed by a build-up phase (escalating peanut doses every 2 weeks, achieving a maintenance dose by 36 weeks). Thereafter, subjects are on a maximally tolerated maintenance dose (165 mcg to 3,696 mcg) for >= 8 weeks. After 44 weeks of open label SLIT, subjects are given a 5,000 mg Oral Food Challenge (OFC) using peanut powder. SLIT=Sublingual Immunotherapy
- Low Dose Peanut SLIT (Double Blind to Open Label): After completion of the 5,000 mg Oral Food Challenge (OFC) at Week 44, subjects/study staff are unblinded and subjects continue on an open label peanut protein maintenance dose of 1,386 mcg/day or may attempt escalation up to this dose. Subjects who at their Week 116 Oral Food Challenge (OFC) are not able to consume at least 5,000 mg of peanut powder or 10-fold the amount of peanut powder compared to their baseline OFC will discontinue study therapy. SLIT=Sublingual Immunotherapy
- Placebo (DB) Crossed Over to High Dose Peanut SLIT (OL): After 44 weeks of open label therapy, subjects are given a 5,000 mg Oral Food Challenge (OFC) using peanut powder. After completion of this Week 44 OFC, subjects then either continue on their peanut protein maintenance dose of 3,696 mcg per day or are allowed to attempt escalation up to this dose. Subjects who at their Week 116 Oral Food Challenge (OFC) are not able to consume at least 5,000 mg of peanut powder or 10-fold the amount of peanut powder compared to their baseline OFC will discontinue study therapy. SLIT=Sublingual Immunotherapy
Arm/Group | Low Dose Peanut SLIT Before Week 44 OFC (Double Blind) | Placebo Before Week 44 OFC (Double Blind) | High Dose Peanut SLIT Crossover Before Wk44 Crossover OFC (OL) | Low Dose Peanut SLIT (Double Blind to Open Label) | Placebo (DB) Crossed Over to High Dose Peanut SLIT (OL)
Serious Adverse Events (participants affected / at risk) | 1/20 | 0/20 | 0/17 | 1/18 | 0/17
Other Adverse Events (participants affected / at risk) | 19/20 | 20/20 | 17/17 | 17/18 | 15/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose Peanut SLIT Before Week 44 OFC (Double Blind) (N=20) | Placebo Before Week 44 OFC (Double Blind) (N=20) | High Dose Peanut SLIT Crossover Before Wk44 Crossover OFC (OL) (N=17) | Low Dose Peanut SLIT (Double Blind to Open Label) (N=18) | Placebo (DB) Crossed Over to High Dose Peanut SLIT (OL) (N=17)
Anaphylactic Reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Low Dose Peanut SLIT Before Week 44 OFC (Double Blind) (N=20) | Placebo Before Week 44 OFC (Double Blind) (N=20) | High Dose Peanut SLIT Crossover Before Wk44 Crossover OFC (OL) (N=17) | Low Dose Peanut SLIT (Double Blind to Open Label) (N=18) | Placebo (DB) Crossed Over to High Dose Peanut SLIT (OL) (N=17)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear pruritus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (114) | 0 (0) | 1/14 (4)
External ear inflammation (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Conjunctivitis allergic (Eye disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye pruritus (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1/14 (5)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 7 (53) | 1 (1) | 6 (33) | 2 (7) | 2/14 (16)
Abdominal pain (Gastrointestinal disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0/14 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (11)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0/14 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Food Poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (10) | 0 (0) | 1 (1) | 0 (0) | 1/14 (1)
Oral disorder (Gastrointestinal disorders) | 17 (2171) | 6 (23) | 16 (1579) | 14 (1913) | 8/14 (1326)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Swollen tongue (Gastrointestinal disorders) | 3 (8) | 0 (0) | 1 (1) | 0 (0) | 0/14 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0/14 (0)
Chills (General disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 0/14 (0)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0/14 (0)
Influenza like illness (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 1 (2) | 2 (2) | 1 (3)
Allergy to animal (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Chronic sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infectious mononucleosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Kidney infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Meningitis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 4 (6) | 5 (7) | 3 (7) | 3 (4) | 1 (1)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Otitis media (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 4 (5) | 2 (2) | 3 (4) | 3 (3) | 4 (7)
Tinea pedis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 4 (5) | 4 (8) | 3 (6) | 3 (10) | 3 (8)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cartilage injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Ligament injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
Lip injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sports injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Muskuloskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (5)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0/14 (0)
Headache (Nervous system disorders) | 2 (4) | 3 (5) | 3 (6) | 2 (6) | 2 (20)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Sinus headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alcoholism (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1/14 (3)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (3) | 2 (2) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (65) | 0 (0) | 0 (0) | 1 (4) | 1/14 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (4) | 0 (0) | 1 (1) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 (8) | 1 (1) | 2 (4) | 0 (0) | 1/14 (1)
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 9 (51) | 3 (4) | 6 (20) | 3 (56) | 1/14 (259)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (3) | 1 (1) | 1 (2) | 1 (1)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (3) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 2 (5) | 1 (1) | 3 (7) | 0 (0) | 3/14 (7)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0/14 (0)
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0/14 (0)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0/14 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0/14 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 7 (62) | 3 (7) | 2 (2) | 1 (2) | 2/14 (3)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0/14 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 7 (24) | 1 (2) | 6 (34) | 5 (7) | 3/14 (15)
Labial frenectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal septal operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Papilloma excision (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Shoulder operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tonsillectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wisdom teeth removal (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0/14 (0)

LIMITATIONS AND CAVEATS:
Refer to the original results published in the Journal of Allergy and Clinical Immunology, Vol 135, Number 5, page 1247 for a full description of the limitations of the current study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No